CLINICAL TRIAL: NCT07155746
Title: Effect of Simulated Weight Loss on the Energy Cost of Locomotion in Overweight or Obese Adolescents
Acronym: DELOAD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Emile Roux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RIPH2_GADEA_DELOAD; 2025-A01209-40 (Other: ID-RCB)
Record Dates: First submitted 2025-08-19; First posted 2025-09-04 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Obesity and Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescents aged 12 to 16 with obesity defined as a BMI above the 97th percentile (Other): 3 different walking exercises
  Interventions: Other: Incremental walking exercise on an AlterG treadmill (anti-gravity)

INTERVENTIONS:
Other: Incremental walking exercise on an AlterG treadmill (anti-gravity) — One visit with their current weight (BW) One visit with simulated weight loss in adolescents to determine their normal weight (NW-SBW) One visit with simulated weight loss in adolescents to determine their overweight status (OW-SBW).

SUMMARY:
Current literature suggests that part of the energy response to weight loss is not due to changes in fat mass and lean mass, but rather to a homeostatic adaptation aimed at limiting or even preventing weight loss and preserving individuals' energy reserves, an adaptation known as "adaptive thermogenesis". This phenomenon calls for a closer look at the respective contributions of metabolic and mechanical changes induced by weight variations, with greater consideration given to the recently proposed hypothesis of dual regulation of homeostatic energy balance involving both leptin-dependent and "gravitostatic" pathways . While leptin-dependent regulation of body weight has been described and reinforced several times since the 1950s, the gravitostatic conception of this regulation is more recent and hypothesizes that terrestrial animals use gravity to regulate their body weight through receptors and pathways that have not yet been identified. This regulation would involve adaptations in energy consumption based on body weight when working against gravity, involving weight detection by osteocytes in weight-bearing bones, and leading to feedback regulation of energy metabolism and body weight . Preclinical and clinical studies conducted on rodents and human participants have shown a reduction in body weight after several weeks of mechanical overload (simulating weight gain), explained by adaptations in their food intake and energy metabolism , adaptations suggested to be particularly due to the regulation of muscle mass. Interestingly, preliminary results from this group highlight specific post-weight loss energy adaptations to such simulated weight regain in adolescents with obesity, suggesting the establishment of specific mechanisms promoting weight regain. Indeed, after weight loss, energy metabolism during locomotion was explored with and without simulated weight regain, and interestingly, energy expenditure did not return to pre-weight loss values, as a potential means of preserving weight regain. More recently, the investigators team has been able to show that such mechanical simulation of weight gain in adolescents with obesity but stable weight does not lead to an increase in their energy expenditure during locomotion, further reinforcing a susceptibility to not activating energy defense mechanisms against this weight gain.Overall, these results suggest the presence of mechanisms for preserving body mass by conserving energy stores as a compensatory defense system against weight loss, while highlighting the absence of activation of these mechanisms in the context of simulated weight gain. Indeed, while the compensatory mechanisms implicated in response to weight fluctuations have thus far been nutritional in nature, these energy adaptations, if confirmed, would suggest an upstream activation mechanism, particularly as a tonic signal for homeostatic control.

It seems necessary to study in greater depth the energy adaptations to weight variations in young people with obesity, both metabolic and mechanical, in order to better understand the control of their energy balance and the mechanisms involved, which corresponds to the objectives of this project.

The objective of this project is therefore to study energy adaptations (energy cost and use of energy substrates) to simulated weight loss during incremental walking exercise. Adolescents with obesity will perform a walking exercise on an AlterG (anti-gravity) treadmill, first without and then with a simulated weight loss that places them in the overweight or normal weight category.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12 to 16 (inclusive), at Tanner stage 3-5, with obesity defined as a body mass index (BMI) above the 97th percentile according to national growth charts.
* No regular consumption of tobacco or alcohol,
* No diet (no calorie restriction, no specific diet such as a normal-calorie diet enriched with protein, vegetarian, or other),
* Adolescents affiliated with the social security system or equivalent,
* Adolescent who has been informed and has given written consent to participate in the study,
* Signed consent of both holders of parental authority (or one in the event of death, major incapacity, or withdrawal of parental authority).

Exclusion Criteria:

* Refusal to participate in the study,
* Refusal of consent by parents or guardians,
* Participation in regular and intense physical and sporting activities (no more than 150 minutes of moderate structured activity per week (according to WHO recommendations),
* Medical or surgical history deemed by the investigator to be incompatible with the study,
* Presence of diabetes or any other condition limiting the application of either strategy being tested,
* Adolescents undergoing energy restriction or a weight loss program through physical activity at the time of inclusion or during the previous 6 months,
* Taking medications that may interfere with the study results.
* Adolescents with cardiovascular problems, i.e., subjects with a history of cardiovascular and/or neurovascular disease, as well as subjects with cardiovascular and/or neurovascular risk factors (excluding obesity/overweight).
* Surgery in the previous 3 months,
* Adolescents who are currently excluded from another study,
* Pregnant or breastfeeding adolescents,
* Adolescents under guardianship/curatorship or legal protection,
* Parents under guardianship/curatorship or legal protection.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-09-12 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Energy expenditure during incremental walking exercise measured by portable calorimetry | 3 Months
  Energy expenditure will be assessed during walking exercise using portable indirect calorimetry (MetaMax, Inc.).
  Indirect calorimetry is one of the classic methods for measuring resting energy expenditure. The contribution of lipid and carbohydrate oxidation will be calculated indirectly by monitoring oxygen consumption and CO2 output according to double unknown equations, assuming that protein oxidation is stable and around 15%.

SECONDARY OUTCOMES:
The use of energy substrates during incremental walking exercise | 3 months
  Energy substrates will be assessed during walking exercise using portable indirect calorimetry (MetaMax, Inc.).
  Indirect calorimetry is one of the classic methods for measuring resting energy expenditure . The contribution of lipid and carbohydrate oxidation will be calculated indirectly by monitoring oxygen consumption and CO2 output using double unknown equations, assuming that protein oxidation is stable and in the order of 15%.
Perception of effort during incremental walking exercise (Borg scale) | 3 months
  At the end of each stage, during the incremental submaximal walking exercise, the adolescents' perception of effort will be assessed using a Borg scale. This scale consists of progressive stages from 6 to 20; 6 corresponds to a perception of very low effort, while 20 corresponds to an effort that is too intense, requiring the exercise to be stopped.

CONTACTS AND LOCATIONS:
Overall Officials: David THIVEL Director of AME2P Laboratory - CLERMONT-FERRAND University, Principal Investigator — Laboratoire des Adaptations Métaboliques à l'Exercice en conditions Physiologiques et Pathologiques